CLINICAL TRIAL: NCT05136872
Title: Continuous Observations of Behavioural Risk Factors in Asia (COBRA)
Acronym: COBRA
Status: Completed | Type: Observational
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Rob M van Dam, Professor, National University of Singapore
Other Study IDs: NUS-IRB-2020-50
Record Dates: First submitted 2021-11-14; First posted 2021-11-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Health Behavior; Diet, Healthy; Physical Activity; Sedentary Behavior; Sleep
Keywords: health behavior; physical activity; sedentary; sleep; eating behavior; GPS; glycaemic response
MeSH Terms: conditions — Health Behavior; Motor Activity; Sedentary Behavior; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to advance understanding of behavioural risk factors for cardiovascular disease and type 2 diabetes in Singapore.

DETAILED DESCRIPTION:
BACKGROUND: Modifiable risk factors for non-communicable diseases, including unhealthy diets and movement behaviours, are influenced by complex and dynamic interactions between people and their social and physical environment. Therefore, understanding patterns and determinants of these risk factors as they occur in real-life is essential to enable the design of precision public health interventions.

AIMS: The aims of this study are to (1) examine patterns of dietary and movement behaviours in real-time as people go about their daily lives, (2) examine how interactions with the social and physical environment influence dietary and movement behaviours, and (3) examine how these patterns differ by ethnicity and other socio-demographic characteristics.

METHOD: This is an observational study in free-living participants over 10 consecutive days, with a 9-day follow-up 6 months later. 1500 participants will be recruited from a large prospective cohort study. Real-time data capture strategies will be used: an ecological momentary assessment (EMA) app with global positioning system (GPS) enabled to collect location data, accelerometers to measure movement, and wearable sensors to monitor blood glucose levels. Participants receive six EMA prompts per day to capture information on diet and movement behaviours (physical activity, sedentary behaviour, sleep), and related contextual factors. A second wave of EMA prompts and GPS monitoring will occur 6 months later. Data will be integrated and analysed using generalised linear models to examine associations between behavioural risk factors and contextual determinants.

ELIGIBILITY:
Inclusion criteria:

* aged 21 to 69 years of age
* citizen or permanent resident of Singapore
* of Chinese, Malay, or Indian ethnicity
* able to read English
* own or have continued access to a smartphone with a data plan
* able to use smartphone apps
* able to walk independently

Exclusion criteria:

* history of stroke, heart disease, renal failure, diabetes mellitus, thyroid disease, cancer, or a serious mental health condition (e.g., schizophrenia, depression, or dementia)
* have had vascular bypass surgery or angioplasty procedure performed
* known sensitivity to medical-grade adhesives
* bleeding disorder

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults in Singapore
Sampling Method: Non-Probability Sample
Enrollment: 1361 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Movement behaviours | continuously for 9 days.
  Movement behaviours (i.e., physical activity, sedentary behaviour, sleep) are measured using a wrist-worn accelerometer.
Glucose concentrations | in 15-minute intervals over 9 days.
  Glucose concentrations are measured using a continuous glucose monitor sensor.
Self-reported food intake | Change in self-reported food intake over time. Data will be collected at 2.5-hour intervals between 8am and 9.30pm over a period of 9 days, and repeated at the 6-month follow-up
  Self-reported food intake measurement through entering of food items and the social and physical environment of eating via an Ecological Momentary Assessment (EMA) smartphone app.
Self-reported movement behaviours | Change in self-reported movement behaviours over time. Data will be collected at 2.5-hour intervals between 8am and 9.30pm over a period of 9 days, and repeated at the 6-month follow-up
  Self-reported movement behaviours (i.e., physical activity, sedentary behaviour, sleep) through entering of the type and social and physical environment context of activity via an Ecological Momentary Assessment (EMA) smartphone app.
Self-reported screen time | Change in self-reported screen time over time. Data will be collected at 2.5-hour intervals between 8am and 9.30pm over a period of 9 days, and repeated at the 6-month follow-up
  Self-reported screen time through entering of the type of screen used and the purpose and the duration of screen time via an Ecological Momentary Assessment (EMA) smartphone app.

SECONDARY OUTCOMES:
Self-reported stress levels | Data will be collected 6 times per day for 9 days, and repeated at the 6-month follow-up.
  Self-reported stress level will be assessed via an Ecological Momentary Assessment (EMA) smartphone app.
Self-reported fatigue | Data will be collected 6 times per day for 9 days, and repeated at the 6-month follow-up.
  Self-reported fatigue will be assessed via an Ecological Momentary Assessment (EMA) smartphone app.
Self-reported positive affect | Data will be collected 6 times per day for 9 days, and repeated at the 6-month follow-up.
  Self-reported positive affect will be assessed via an Ecological Momentary Assessment (EMA) smartphone app.
Self-reported hunger | Data will be collected 6 times per day for 9 days, and repeated at the 6-month follow-up.
  Self-reported hunger will be assessed via an Ecological Momentary Assessment (EMA) smartphone app.

CONTACTS AND LOCATIONS:
Overall Officials: Rob M van Dam, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Saw Swee Hock School of Public Health, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edney SM, Park SH, Tan L, Chua XH, Dickens BSL, Rebello SA, Petrunoff N, Muller AM, Tan CS, Muller-Riemenschneider F, van Dam RM. Advancing understanding of dietary and movement behaviours in an Asian population through real-time monitoring: Protocol of the Continuous Observations of Behavioural Risk Factors in Asia study (COBRA). Digit Health. 2022 Jun 30;8:20552076221110534. doi: 10.1177/20552076221110534. eCollection 2022 Jan-Dec. PMID 35795338